CLINICAL TRIAL: NCT01241357
Title: High-Tc Susceptometer to Monitor Transfusional Iron Overload (NSR Device)
Brief Title: High-Tc Susceptometer to Monitor Transfusional Iron Overload
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Gary M Brittenham, MD, James A. Wolff Professor of Pediatrics, Columbia University
Other Study IDs: AAAE5051; R01FD003702 (FDA)
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Transfusional Iron Overload; Thalassemia Major; Sickle Cell Disease; Myelodysplastic Syndromes; Aplastic Anemia
Keywords: Iron; Iron overload; Hepatic iron concentration; High-temperature superconductivity; Magnetic susceptibility; Susceptometer
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Myelodysplastic Syndromes; Anemia, Aplastic; Iron Overload

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation only: This study has a single arm and no intervention.
  Interventions: Device: Hepatic biomagnetic susceptibility measurement

INTERVENTIONS:
Device: Hepatic biomagnetic susceptibility measurement — Subjects will first have an ultrasound study to determine the location of the liver and measure the distance from skin surface to the liver. Subjects will then be examined with the high Tc susceptometer to determine the amount of iron in the liver. The entire procedure will usually take one-half hour or less.
  Other Names: Hepatic magnetic susceptibility measurement; Superconducting biosusceptometry

SUMMARY:
The proposed research project will continue the application and development of a new method (biomagnetic susceptometry) that measures magnetic fields to determine how much iron is in the liver. The amount of iron in the liver is the best indicator of the amount of iron in the whole body. Measuring the amount of iron in the body is important because either too much (iron overload) or too little iron (iron deficiency) can be harmful. At present, the most reliable way to measure the amount of iron in the liver is to remove a sample of the liver by biopsy, either by surgery or by using a needle which pierces the skin and liver. Iron stored in the liver can be magnetized to a small degree when placed in a magnetic field. In patients with iron overload, the investigators previous studies have shown that magnetic measurements of liver iron in patients with iron overload are quantitatively equivalent to biochemical determinations on tissue obtained by biopsy. In the past the investigators have developed a device to measure the amount of magnetization, which was called a SQUID (Superconducting QUantum Interference Device) susceptometer. This device was validated and in use for over 20 years. The safety, ease, rapidity and comfort of magnetic measurements make frequent, serial studies technically feasible and practically acceptable to patients. The investigators have now developed a new susceptometer, which uses very similar technology to the SQUID, but the investigators believe is more accurate and precise. This study aims to validate this new instrument. The investigators will do prospective, serial studies of the diagnosis and management of patients with iron overload, including thalassemia major (Cooley's anemia), sickle cell disease, aplastic anemia, myelodysplasia, hereditary hemochromatosis, and other disorders. Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
This project will validate our new high-transition-temperature (high-Tc; operating at 77°K, cooled by liquid nitrogen) superconducting magnetic susceptometer as the most clinically effective means for monitoring iron overload in patients who require chronic red blood cell transfusion. Transfusional iron overload is an orphan disease that develops in patients who require regular blood transfusions for treatment of a variety of refractory anemias that are themselves orphan disorders, including sickle-cell disease, thalassemia major (Cooley's anemia), Diamond-Blackfan anemia, aplastic anemia, pure red cell aplasia, hypoplastic and myelodysplastic disorders. In the United States, the number of anemic patients with transfusional iron overload is estimated to be less than 50,000. Without iron-chelating therapy, potentially lethal amounts of iron accumulate in these patients. Because the body lacks an effective means to eliminate excess iron, the iron contained in transfused red cells is progressively deposited in the liver, heart, pancreas and other organs. Cirrhosis, heart failure, diabetes and other disorders develop. Treatment with a chelating agent capable of sequestering iron and permitting its excretion from the body provides a means of managing transfusional iron overload that can prolong survival and avert or ameliorate iron-induced organ damage. Two iron-chelating agents are now approved for use in the U.S. for the treatment of transfusional iron overload: (1) deferoxamine B (Desferal®), a parenteral agent in use for almost four decades, and (ii) deferasirox (Exjade®), an orally administered agent introduced in 2005. With both chelators, optimal management of patients requires careful monitoring of body iron to prevent iron-induced toxicity while avoiding adverse effects of excessive chelator administration. Our laboratories originally proposed that storage iron (ferritin and hemosiderin) could be non-invasively assessed in vivo by measurement of magnetic susceptibility. We subsequently developed low-transition-temperature (low-Tc; operating at 4°K, cooled by liquid helium) superconducting quantum interference device (SQUID) susceptometry as a clinical method for quantitation of hepatic iron stores. The transition temperature is the temperature at which the electrical resistance of a superconducting material drops to zero. The safety, ease, rapidity and comfort of magnetic measurements have made frequent, serial investigations technically feasible and practically acceptable to patients. Susceptometry permits accurate, direct, reliable, and repeated measurements of hepatic iron stores. Despite these advantages, the cost (about $1,000,000 per device), instrumental complexity and need for liquid-helium cooling of the low-Tc susceptometers restricted clinical adoption of the method. Worldwide, only four low-Tc susceptometers have been used clinically (in New York, Oakland, Hamburg and Turin). Recently, with the support of a Bioengineering Research Partnership Grant (R01 DK057209), we have made a series of technological breakthroughs and instrumental innovations that have made possible replacement, redesign and refinement of the elements of the low-Tc susceptometer, operating at 4°K in liquid helium, with components able to function at 77°K in liquid nitrogen. This new high-Tc susceptometer, the first medical device utilizing the phenomenon of high-temperature superconductivity, is an inexpensive instrument that can easily be used in a hospital environment. These Phase 2 clinical studies are designed to test the hypothesis that measurements of hepatic iron stores with our new high-Tc susceptometer are clinically superior to all other available methods and to supply essential data needed for FDA approval of the medical device. The proposed project has three specific aims:

1. to calibrate the high-Tc susceptometer with the results of biochemical analysis of tissue from liver explants from adult and pediatric patients undergoing liver transplantation and from clinically indicated liver biopsy; and
2. to prospectively validate the high-Tc susceptometer using the results of biochemical analysis of tissue from liver explants from adult and pediatric patients undergoing liver transplantation and from clinically indicated liver biopsy; and
3. to prospectively compare measurements of hepatic iron concentration by the high-Tc susceptometer with (i) estimates derived from liver magnetic resonance imaging (MRI) relaxation rates (R2, R2*, signal intensity ratios), (ii) with determinations of serum ferritin, and (iii) with histopathological examination, using biochemical analysis of liver storage iron concentrations as the reference standard.

FDA approval of an affordable, readily usable instrument for the non-invasive measurement of hepatic iron stores would lead to major advances in the management of patients with transfusional iron overload that would find immediate and widespread clinical use both in the U.S. and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* being an adult male, nonpregnant female or child who is scheduled for liver transplantation, has transfusional iron overload or is healthy with no known disorder affecting body iron stores,
* being of sufficient size for the susceptometer (about 15 kg body weight),
* being able to lie quietly during the measurement procedure (about 5 to 10 minutes),
* being either able to give fully informed consent or, if a minor, with a parent or legal guardian who is able to give fully informed consent for participation of the minor.

Exclusion Criteria:

* any form of magnetic contamination or electrical device which cannot be removed for the magnetic measurement procedure, including jewelry, pacemakers, artificial joints, metal staples, indwelling catheters with metallic components, dental braces or other magnetic objects;
* obesity, ascites or other conditions in which the liver to surface distance exceeds 25 mm;
* pregnancy, treatment for mental illness, imprisonment, institutionalization, or any condition that impairs ability to provide fully informed consent.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants who are eligible for this study include: (i) patients scheduled for clinically indicated liver transplantation or liver biopsy, (ii) patients with transfusional iron overload followed in adult and pediatric hematology, and (iii) healthy individuals participating as control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hepatic non-heme iron concentration determined by biomagnetic susceptometry | 2 years
  The primary study analysis will be a comparison of the results of measurements of the hepatic storage iron concentration by biomagnetic susceptometry with the results of biochemical analysis of the storage iron concentration in liver tissue.

SECONDARY OUTCOMES:
Serum ferritin concentration | 2 years
  A secondary study analysis will be a comparison of the results of measurements of the hepatic storage iron concentration by biomagnetic susceptometry with the results of measurements of the serum ferritin concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Gary M. Brittenham, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Farrell DE, Allen CJ, Whilden MW, Kidane TK, Baig TN, Tripp JH, Brown RW, Sheth A, Brittenham GM. A new instrument designed to measure the magnetic susceptibility of human liver tissue in vivo. IEEE Trans Magnetics 2007;43:3543-3554.
- [Background] Farrell DE, Allen CJ, Whilden MW, Tripp JH, Usoskin A, Sheth A, Brittenham GM. Magnetic measurement of liver iron stores: engineering aspects of a new scanning susceptometer based on high temperature superconductivity. IEEE Trans Magnetics 2007; 43:4030-4036.